CLINICAL TRIAL: NCT03763682
Title: A Multicentre, Prospective, Open-label, 2 Groups Study to Assess the Safety and Performance of the Genio™ Bilateral Hypoglossal Nerve Stimulation System for the Treatment of Obstructive Sleep Apnoea in Adult Patients With and Without Complete Concentric Collapse of the Soft Palate
Brief Title: BilatEral Hypoglossal Nerve StimulaTion for TreatmEnt of ObstRuctive SLEEP Apnoea With and Without Complete Concentric Collapse
Acronym: BETTER SLEEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to operational challenges impacting protocol execution across sites.
Sponsor: Nyxoah S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BETTER SLEEP
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: prospective, open-label, 2 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genio(TM) system therapy (Experimental): Genio(TM) bilateral hypoglossal nerve stimulation system
  Interventions: Device: Genio(TM) bilateral hypoglossal nerve stimulation system

INTERVENTIONS:
Device: Genio(TM) bilateral hypoglossal nerve stimulation system — Subjects will be consented, enrolled and eligibility criteria checked. If the subject is eligible, subject will proceed with the Genio(TM) implant implantation. Six (6) weeks after implantation, the implant will be activated and the subject will be assessed at 1 month plus 1 week, 2, 3, 4, 5 and 6 month(s) after implantation

SUMMARY:
The objective of this study is to explore the safety and performance of the Genio™ system in adult obstructive sleep apnoea (OSA) patients with and without complete concentric collapse of the soft palate over a period of 4.5 months of treatment (i.e. 6 months post-surgery) measured by the AHI, at rest to determine if there is a difference in performance between the two populations.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentric, 2 groups study to assess the safety and performance of the Genio™ system in adult obstructive sleep apnoea (OSA) patients with and without complete concentric collapse of the soft palate. Participants will be consented, enrolled and eligibility criteria checked. If the participant is eligible, participant will proceed with the Genio™ IS implantation. Six (6) weeks after implantation, the implant will be activated and study visits will be scheduled at Week 7, Month 2, Month 3, Month 4, Month 5 and Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 21 and 75 years of age
* Body mass index (BMI) ≤ 32 kg/m2
* Obstructive apnoea-hypopnea index (AHI) of 15-50 events/hour
* Participants who have either not tolerated, have failed or refused positive airway pressure (PAP) treatments.

Exclusion Criteria:

* Unable or incapable of providing informed written consent
* Unwilling or incapable of returning to all follow-up visits and sleep studies, including evaluation procedures and filling out questionnaires

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence of serious device-related adverse events recorded during the study | 6 months
Change from baseline to 6 months post implantation in the apnoea-hypopnea index (AHI) | Change from baseline to 6 months post implantation in the apnoea-hypopnea index (AHI)

SECONDARY OUTCOMES:
Change from baseline to 6, 12, 24 and 36 months post implantation in Oxygen Desaturation Index (ODI) | 6,12, 24, 36 months
Change from baseline to 12, 24 and 36 months post implantation in Apnea Hypopnea Index (AHI) | 12, 24, 36 months

OTHER OUTCOMES:
Therapy response rate | 6, 12, 24, 36 months
  Response is defined as a reduction in AHI from baseline to 6 months of 50% or higher and apnoea-hypopnea index (AHI) at 6 months less than 20.
Sleep-related quality of life, measured by functional Outcomes of Sleep Questionnaire (FOSQ-10) score | 6, 12, 24, 36 months
  The questionnaire assesses the impact of excessive sleepiness on functional outcomes relevant to daily behaviors and sleep-related quality of life. It uses a 4-point Likert response format (1= extreme difficulty to 4=no difficulty) for 5 subscales: 1) activity level (3 items), 2) vigilance(3 items), 3) intimacy and sexual relationships (1 item), 4) general productivity (2 items), and 5) social outcomes (1 item). A total score is calculated and an increase is considered an improvement.
Change from baseline to 6 months post implantation in daytime sleepiness measured with Epworth Sleepiness Scale (ESS) | 6, 12, 24, 36 months
  The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives. The scores for the eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought. A reduction in ESS is considered a better outcome with a decrease of 2 points considered to be clinically significant.
Change from baseline to 6 months post implantation in snoring intensity | 6, 12, 24, 36 months
  Measured subjectively by the bed partner using a 5 point scale of no scoring, light snoring, medium snoring, very loud snoring, to leaving the bedroom.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Westmead Private Hospital, Westmead, New South Wales
  - Wollongong Private Hospital, Wollongong, New South Wales
  - Institute Breathing and Sleep Austin Hospital, Heidelberg, Victoria
  - Hollywood Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No